CLINICAL TRIAL: NCT01645150
Title: Pilot Study on the Effects of Strength Training on Cancer Related Fatigue in Cancer Patients During Tyrosine Kinase Inhibitor Therapy
Brief Title: Reduction of Cancer Related Fatigue in Patients During TKI Therapy
Acronym: RECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-154/2012
Record Dates: First submitted 2012-06-11; First posted 2012-07-20 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: All Tumor Entities Treated With TKI Therapy
Keywords: physical activity; exercise; training; fatigue; cancer; TKI; tyrosine kinase inhibitor
MeSH Terms: conditions — Motor Activity; Fatigue; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strength training group (Experimental): 12 weeks of progressive strength training
  Interventions: Behavioral: Progressive strength training
- Control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Progressive strength training — 12 weeks of supervised progressive strength training
  Arms: Strength training group

SUMMARY:
The purpose of this pilot study is to determine the effects of a 12-week resistance training program on cancer related fatigue in cancer patients receiving tyrosine kinase inhibitor (TKI) therapy. It is hypothesized that incidence and severity of cancer related fatigue can be reduced by exercise training in this population which leads to an improved treatment completion rate.

ELIGIBILITY:
Inclusion Criteria:

* Male and female cancer patients
* Prior to tyrosine kinase inhibitor therapy (any substance, any line)
* Age: at least 18 yrs
* Body mass index (BMI): at least 18 kg/m2
* ECOG performance status: at most 2
* Must be able to meet the requirements of the study protocol

Exclusion Criteria:

* Acute infectious diseases
* No ambulatory ability
* Severe neurological disorders
* Severe cardiovascular diseases
* Severe pulmonary insufficiency
* Severe renal insufficiency
* Other current tumor diseases
* Conditions rendering compliance impossible
* Participation in regular strength training

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in cancer related fatigue | From baseline to the 6th and 12th week of training.
  Assessed via the Multidimensional Fatigue Inventory (MFI).

SECONDARY OUTCOMES:
Change in muscle strength of the knee extensor, hip flexor and forearm flexor muscles. | From baseline to the 12th week of training.
  Assessed isokinetically and isometrically via an IsoMed2000 test system.
Change in endurance capacity | From baseline to the 12th week of training.
  Maximal oxygen uptake (VO2max) assessed in a maximal incremental cycling test.
Change in body composition | From baseline to the 12th week of training
  Assessed via bio-impedance measurement.
Change in quality of life | From baseline to the 6th and 12th week of training.
  Assessed via the EORTC QLQ C30.
Change in depression | From baseline to the 6th and 12th week of training.
  Assessed via "Allgemeine Depressionsskala" (ADS).
Time of the first tumor progression under TKI therapy | Within the first 6 months of TKI therapy
Time of reduction or replacement of TKI therapy | Within the first 6 months of TKI therapy

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Grüllich, MD, Principal Investigator — National Center for Tumor Diseases Heidelberg (GermanCRC/University Hospital Heidelberg) Germany; Friederike Scharhag-Rosenberger, PhD, Principal Investigator — National Center for Tumor Diseases Heidelberg (GermanCRC/University Hospital Heidelberg) Germany; Joachim Wiskamann, PhD, Principal Investigator — National Center for Tumor Diseases Heidelberg (GermanCRC/University Hospital Heidelberg) Germany; Dirk Jäger, Professor, Study Chair — National Center for Tumor Diseases Heidelberg (GermanCRC/University Hospital Heidelberg) Germany; Karen Steindorf, Professor, Study Chair — National Center for Tumor Diseases Heidelberg (GermanCRC/University Hospital Heidelberg) Germany
Locations (1):
- National Center for Tumor Diseases Heidelberg (German Cancer Research Center/University Hospital Heidelberg), Heidelberg, Germany

REFERENCES:
- [Derived] Rosenberger F, Wiskemann J, Vallet S, Haag GM, Schembri E, Jager D, Grullich C. Resistance training as supportive measure in advanced cancer patients undergoing TKI therapy-a controlled feasibility trial. Support Care Cancer. 2017 Dec;25(12):3655-3664. doi: 10.1007/s00520-017-3788-3. Epub 2017 Jun 30. PMID 28667563